CLINICAL TRIAL: NCT01661569
Title: A Randomised Controlled Trial to Investigate the Effects of the Headspace Mindfulness Smartphone App on Psychological Well-being and Biological Indicators of Stress in the Workplace
Brief Title: A Randomised Controlled Trial to Investigate the Effects of a Mindfulness Smartphone App on Well-being in the Workplace
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University College, London (Other)
Collaborators: British Heart Foundation (Other); Headspace Meditation Limited (Industry); Technical University Dresden (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3035/002
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Well-being, Work Stress
Keywords: Mindfulness; meditation; stress; well-being; work stress; blood pressure; cortisol
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Headspace On-the-go app (Experimental): Participants were given access to a 45-day mindfulness meditation programme via the Headspace smartphone app
  Interventions: Other: Headspace On-the-go app
- Waitlist control (No Intervention): Participants will be asked to wait for 8 weeks before starting the intervention

INTERVENTIONS:
Other: Headspace On-the-go app — Participants will be given access to a 45-day programme of mindfulness meditation, created and branded by Headspace. They will be encouraged to listen to one meditation podcast each day, or as frequently as possible over 8 weeks.
  Other Names: Mindfulness meditation smartphone app
  Arms: Headspace On-the-go app

SUMMARY:
We propose a randomised controlled trial in a workplace setting to investigate whether a smartphone-delivered programme of mindfulness meditation influences psychological and biological indicators of well-being.

We hypothesise that after 8 weeks participants who complete the meditation programme will show increases in psychological well-being and reduced activation of stress-related biological pathways.

DETAILED DESCRIPTION:
Mindfulness-based therapies can reduce depressive symptoms in patients and healthy subjects. Therapies such as MBSR (mindfulness-based stress reduction) typically consist of 8 group sessions led by an experienced practitioner, plus home practice and one full day of meditation. In this study we aim to investigate whether a mindfulness programme delivered as a series of podcasts on a mobile phone app could lead to gains in well-being and a reduction in stress.

ELIGIBILITY:
Inclusion Criteria:

* Employees of a UK high-tech company
* Raised levels of work stress (overcommitment>2) or depression (CESD>1)

Exclusion Criteria:

* treated for anxiety, depression or hypertension
* taking medication containing steroids

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Well-being | 8 weeks
  Psychological well-being will be assessed using the Warwick Edinburgh Mental Well-Being Scale

SECONDARY OUTCOMES:
Blood pressure | 8 weeks
  Blood pressure over the working day will be measured as an indicator of activation of the stress response

OTHER OUTCOMES:
Psychological stress | 8 weeks
  Stress will be measured using the Perceived Stress Scale and measures of job strain, based on Karasek (where job strain is a combination of high demands and low control).
Cortisol | 8 weeks
  Hair cortisol concentration, as an indicator of activation of the HPA axis

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Steptoe, DPhil, DSc, FMedSci, Principal Investigator — University College, London
Locations (1):
- UK high-tech company office, London, United Kingdom